CLINICAL TRIAL: NCT02548572
Title: Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa - a Safety and Efficacy NSR Device Study - A Multicenter Study
Brief Title: Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa - a Safety and Efficacy Multicenter Study
Acronym: TES/RP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit patients
Sponsor: Wills Eye (Other)
Collaborators: Okuvision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMC1TES/RP
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Retinitis Pigmentosa
Keywords: Transcorneal Electrical Stimulation; TES; Retinitis Pigmentosa; RP
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group (Experimental): Subjects in the treatment group will undergo bilateral transcorneal electrical stimulation using OkuStim device once a week for fifty-two weeks
  Interventions: Device: Transcorneal Electrical Stimulation using Okustim device
- Sham group (Placebo Comparator): Subjects in the Sham group will wear the OkuSpex and OkuEl (applied to cornea upon the lower lid) and be attached to the OkuStim device in the same manner as the treatment group, but will receive no electrical stimulation for the 30 minutes that the TES fiber is applied to the cornea (even though the device has been turned on) once a week for fifty-two weeks
  Interventions: Device: Transcorneal Electrical Stimulation using Okustim device

INTERVENTIONS:
Device: Transcorneal Electrical Stimulation using Okustim device — The Okustim® stimulation device is a battery-powered electronic neuro-stimulator, which delivers a weak electrical pulse. This current is delivered to the eyes by the OkuStim® device using the "OkuEl®" electrodes, which are held in place via the "OkuSpex®" frame. In this study the treatment level will be held constant at 0.8 mA for all study subjects. After switching on the neuro-stimulator, the subject's retina will be stimulated through specific electrodes (OkuEl, held in position by the OkuSpex) worn on the face with the predetermined intensity and time period (delivered by the OkuStim device).

SUMMARY:
Several studies have shown that TES in RP patients may help to slow the progressive deterioration of this degenerative disease. The end point of this clinical trial is to slow or stop disease progression with weekly treatment using TES for 1 year.

DETAILED DESCRIPTION:
The following proposed study (ICM1TES/RP) will investigate the therapeutic aspects of transcorneal electrical stimulation (TES) on the eye in patients with retinitis pigmentosa (RP). It will utilize the Okuvision TES system, a Wills Eye Hospital-sponsored FDA non-significant risk (NSR) medical device, OkuStim® (CE-marked OkuStim®) for the application of electrical stimulation directly to the eye via a corneal contact electrode.

Study Design - Multi-center, prospective, randomized sham controlled 1:1 Clinical trial.

Study treatments - Patients will be randomized in a 1:1 ratio. Patients in treatment group will have TES at 200% of phosphene threshold for 30 minutes once weekly for 52 weeks in both eyes. Patients in sham group will also wear electrodes on both eyes, but no energy is turned on and both eyes are sham.

Duration of study - anticipated duration is 36 months, 12 months for recruitment, 12 months for treatment and sham groups and followed for 18 months, plus 6 months for analysis.

Inclusion Criteria - Diagnosis of RP, 22-80 years of age, no other ocular disease, able to complete all visits.

Treatments - TES, 30 minute treatment weekly for 52 weeks at 0.8mA

Number of patients - 90 patients in treatment arm and 90 patients in sham arm. Electrodes will be placed on both eyes, both eyes will be treated in treatment group and in the sham group both eyes will be considered. However due to the possibility of drop out using 15% we will recruit 210 patients (15 patients per center).

Screening -

1. VA & Phosphene threshold evaluation
2. Vfiii4e, vfVe, Octopus 900, complete eye exam, fundus photo, OCT and Contrast sensitivity, electro-physiology.
3. Eligibility requirements met, then schedule baseline.

Tests - Base Line: VA, vfiii4e, vfVe, Octopus 900, complete eye exam, fundus photo, OCT, Contrast sensitivity, NEI VFQ-25, Photopic B-wave ERG, blood draw for genetic test (unless genetic profile has been done).

3 Month visit: VA, eye exam, Phosphene threshold, OCT & Photopic B-wave.

6 Month visit: VA, vfiii4e, vfVe, Octopus 900, complete eye exam, OCT & Contrast sensitivity, phosphine threshold & Photopic B-wave.

9 Month visit: VA, eye exam, Phosphene threshold, OCT & Photopic B-wave.

12 Month visit: VA, vfiii4e, vfVe, Octopus 900, complete eye exam, OCT & Contrast sensitivity, NEI VFQ-25, phosphene threshold & Photopic B-wave

18 Month visit: VA, vfiii4e, vfVe, Octopus 900, complete eye exam, OCT & Contrast sensitivity, NEI VFQ-25 & phosphene threshold & Photopic B-wave.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Retinitis Pigmentosa.
2. Adult patients, 22-80 years of age, having provided written informed consent and HIPAA authorization.
3. LogMAR VA 1.00 or better in both eyes.
4. Octopus 900 Central Visual Field ≥10 degrees diameter around central fixation using stimulus sizes III4e and V4e in both eyes on kinetic testing.
5. Agree to discontinue Vitamin A use and no intake for at least 2 months prior to baseline visit.

Exclusion Criteria:

1. Visual field loss as demonstrated by Octopus 900 kinetic perimetry as <10 deg of remaining central visual field using stimulus sizes III4e and V4e.
2. Due to distance or other reason, patients unable to travel to Philadelphia or respective centers for the treatment procedures and follow-up examinations.
3. Diabetic retinopathy
4. Ocular neovascularisation of any origin
5. After arterial or venous occlusion
6. After retinal detachment or any vitreoretinal surgery with or without implantation.
7. Silicone oil tamponade
8. Dry or exudative age-related macular degeneration
9. Macular edema involving the foveal center as determined by SD-OCT
10. All forms of glaucoma
11. Any form of corneal degeneration that reduces visual acuity
12. Systemic diseases that are difficult to control or manage, which could hinder regular attendance at follow-up examinations
13. Patients in a permanently poor general condition, which could hinder regular attendance at follow-up examinations
14. Patients in whom phosphenes are only inducible at greater than, but not including, 0.8 mA.
15. Forms of mental illness related to the bipolar affective and schizoid-affective disorders, epilepsy, and all forms of dementia
16. Simultaneous participation in another interventional study or history of interventions whose effect may still persist
17. Current pregnancy, or being a woman with childbearing potential who is unwilling to use medically acceptable means of birth control for the study duration, or a woman unwilling to perform a pregnancy test at study entry
18. Any patient can be excluded from the study as determined by the Principal Investigator.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Octopus vfiii4e (Progressive slowing of Visual Field deterioration) | 76 weeks
  Octopus vfiii4e test will be done at Screening visit, Baseline visit, Week 26, Week 53 and Week 76 to analyze progressive slowing of Visual Field deterioration

SECONDARY OUTCOMES:
Visual acuity (VA) | 76 weeks
  VA testing will be done at all visits
Contrast sensitivity | 76 weeks
  Contrast sensitivity testing will be done at Baseline visit, Week 26, Week 53 and Week 76
NEI-VFQ-25 total score & subscores | 53 weeks
  NEI-VFQ-25 survey will be filled out at Baseline visit and at Week 53
Photopic b-wave ERG | 76 weeks
  Photopic b-wave ERG test will be done at Baseline visit, Week 13, Week 26, Week 39, Week 53 and Week 76

OTHER OUTCOMES:
Change in phosphene threshold detection levels | 76 weeks
  Change in phosphene threshold detection levels will be done at Screening visit, Baseline visit, Week 13, Week 26, Week 39, Week 53 and Week 76. This is an exploratory efficacy endpoint.
Octopus GATE (static) | 76 weeks
  Octopus GATE (static) test will be done at Screening visit, Baseline visit, Week 26, Week 53 and Week 76. This is an exploratory efficacy endpoint.
Octopus vf V4e (kinetic) | 76 weeks
  Octopus vf V4e (kinetic) test will be done at Screening visit, Baseline visit, Week 26, Week 53 and Week 76. This is an exploratory efficacy endpoint.
SD-OCT (ez analysis) | 76 weeks
  SD-OCT (ez analysis) test will be done at Screening visit, Baseline visit, Week 26, Week 53 and Week 76. This is an exploratory efficacy endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hyman, PhD, Study Director — Wills Eye Hospital
Locations (1):
- Wills Eye Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes